CLINICAL TRIAL: NCT03858582
Title: A Phase II, Neo-adjuvant Pembrolizumab, Docetaxel, Cisplatin Therapy Followed by Surgery and Pembrolizumab Consolidation Therapy in Locally Advanced Thymic Epithelial Tumor (TET)
Brief Title: neoadjuvant_thymic Epithelial Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Principal Investigator, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-11-105
Record Dates: First submitted 2019-02-14; First posted 2019-02-28 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Thymic Epithelial Tumor
MeSH Terms: conditions — Thymic epithelial tumor | interventions — pembrolizumab; Radiation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Patients with R0 resection will receive pembrolizumab 200mg for 32 cycles.
  Interventions: Drug: pembrolizumab
- Arm B (Experimental): Patient who had R1 resection will receive radiation 52.8Gy/24Fx with pembrolizumab 200mg for 32 cycles. Patients who had R2 resection will receive radiation 59.4Gy/27Fx with pembrolizumab 200mg for 32 cycles.
  Interventions: Drug: pembrolizumab; Radiation: Radiation
- Arm C (Experimental): Patients who showed non-progressive disease (PD) to initial neoadjuvant therapy but remained unresectable will receive radiation 59.4Gy/27Fx with 200mg for 32 cycles.
  Interventions: Drug: pembrolizumab; Radiation: Radiation

INTERVENTIONS:
Drug: pembrolizumab — pembrolizumab 200mg
Radiation: Radiation — 52.8Gy/24Fx or 59.4Gy/27Fx
  Arms: Arm B; Arm C

SUMMARY:
This is a Phase II single center, open-label, single arm study in patients with unresectable thymic epithelial tumors (Masaoka stage III, IVA). Patients will be treated with Pembrolizumab 200 mg, Docetaxel 75mg/m2, Cisplatin 75mg/m2 every 3 weeks for 3 cycles and will be evaluated for the operability. Patients with R0 resection will receive pembrolizumab 200mg for 32 cycles. Patient who had R1 resection will receive radiation 52.8Gy/24Fx with pembrolizumab 200mg for 32 cycles. Patients who had R2 resection will receive radiation 59.4Gy/27Fx with pembrolizumab 200mg for 32 cycles. Patients who showed non-progressive disease (PD) to initial neoadjuvant therapy but remained unresectable will receive radiation 59.4Gy/27Fx with 200mg for 32 cycles. Otherwise patients are off the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 19 years of age on the day of signing informed consent with histologically confirmed diagnosis of TETs will be enrolled in this study.
2. Locally advanced stage (Modified Masaoka stage III or IVa)
3. No previous chemotherapy treatment history
4. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
5. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
6. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
7. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
8. Have measurable disease based on RECIST 1.1.
9. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously treated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
10. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
2. Has received prior systemic anti-cancer therapy including investigational agents except patient had no active treatment for past 5 years.
3. Has received prior radiotherapy.
4. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has a known additional malignancy that is progressing or has required active treatment. Exception include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a known history of Human Immunodeficiency Virus (HIV).
12. Has an active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] positive) infection or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
13. Has a known history of active TB (Bacillus Tuberculosis). Old TB patient can be participated by investigator's decision.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
17. Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension or arrhythmia
18. Has a treatment history wih mAb within 4 weeks prior to the first dose of trial treatment
19. Has a known history of psychosis or substance abuse

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response rate defined by ≤ 10% of tumor composed of viable tumor | about 36months
  Major pathologic response rate defined by ≤ 10% of tumor composed of viable tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bang YH, Noh JM, Lee B, Choi YL, Yang K, Pyo H, Kim H, Kim J, Jung HA, Sun JM, Lee SH, Ahn JS, Ahn MJ, Jeon YJ, Lee J, Cho JH, Kim HK, Choi YS, Park SY, Park S. Perioperative Pembrolizumab for Locally Advanced Thymic Epithelial Tumors: A Single-Arm, Phase 2 Trial. J Thorac Oncol. 2025 Dec;20(12):1829-1842. doi: 10.1016/j.jtho.2025.08.011. Epub 2025 Oct 19. PMID 41109992